CLINICAL TRIAL: NCT07121972
Title: Mirai-MRI: Multi-site Prospective Validation of AI Models for Breast Cancer Risk
Brief Title: Mirai-MRI: Validation of AI Models for Breast Cancer Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25756; NCI-2025-06040 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-08-06; First posted 2025-08-14 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cancer Risk; Breast Cancer Risk
Keywords: Screening; BI-RADS
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Supplemental MRI (Experimental): Participants identified as Mirai high-risk on a negative/benign screening mammogram will receive a supplemental MRI within 12 months of receiving a screening mammogram. Breast cancer risk following the Tyrer-Cuzick risk model will be assessed for comparison.
  Interventions: Procedure: Magnetic resonance imaging (MRI); Device: Artificial Intelligence (AI)

INTERVENTIONS:
Procedure: Magnetic resonance imaging (MRI) — Undergo Magnetic resonance (MR) imaging
  Other Names: MRI; MRI Scan
Device: Artificial Intelligence (AI) — AI applied to MRI images
  Other Names: AI Models; AI Algorithm

SUMMARY:
This is a multi-center, single arm trial to evaluate the cancer detection rate of supplemental screening magnetic resonance imaging (MRI) in participants who are high-risk by Mirai-MRI assessment. Mirai is an accurate cancer risk model based on full-resolution mammograms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the cancer detection rate (CDR) of supplemental screening breast MRI in participants who are high-risk by the Mirai model

SECONDARY OBJECTIVES:

I. To estimate the CDR of supplemental screening breast MRI in participants with high Mirai risk and low (<20%) lifetime Tyrer-Cuzick (TC) risk.

II. To compare the CDR of supplemental screening breast MRI in participants with high Mirai risk and high (≥ 20%) lifetime TC risk versus CDR in participants with high Mirai risk and low (<20%) lifetime TC risk.

III. To estimate the positive predictive value (PPV)1, PPV2, and PPV3 of supplemental MRI screening in participants with high Mirai risk.

IV. To estimate the false positive rate (1 - specificity) of supplemental screening MRI in participants with high Mirai risk.

V. To evaluate the tumor size, stage, grade, histological and molecular subtypes, Ki-67 percentage, and lymph node involvement of cancers detected on supplemental screening MRI in Mirai high risk participants.

VI. To evaluate the association between race/ethnicity, menopausal status, hormonal status, breast density, family history of cancer, and CDR in Mirai high-risk participants.

ELIGIBILITY:
Inclusion Criteria:

1. All asymptomatic participants assigned female at birth, ages 40-89 years old with screening mammography assessed as Breast Imaging Reporting and Data System (BI-RADS) 1, BI-RADS 2, or initial BI-RADS 0 with subsequent diagnostic mammogram assessed as BI-RADS 1 or BI-RADS 2.
2. Screening mammogram assessed as high-risk by Mirai (top 3 percentile of 2-year risk).
3. Availability of a routine screening mammogram report, along with a subsequent diagnostic mammogram report if applicable, and access to the corresponding Digital Imaging and Communications in Medicine (DICOM) images.
4. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Screening mammogram that is assessed as BI-RADS 0 for technical recall.
2. Contraindications for MRI:

   1. Metallic foreign body in the eye.
   2. MRI unsafe implants and/or medical devices.
   3. Adverse reaction to a (gadolinium-based) contrast agent in the past.
   4. Pregnant women.
   5. Claustrophobia.
   6. Exceeds site specific size and/or weight limit for MRI.
3. If the participant meets site-specific criteria for screening estimated glomerular filtration rate (eGFR) prior to MRI, participants with severely impaired renal function (GFR < 30 mL/min) will be excluded. According to University of California, San Francisco's policy for MRI with contrast (gadolinium-containing), serum creatinine with calculation of eGFR should be obtained within 6 weeks of the MRI study for participants with any of the following risk factors:

   1. History of "kidney disease" as an adult, including renal tumor or transplant.
   2. Diabetes treated with insulin or other prescribed medications.
   3. Hypertension (high blood pressure) requiring medication.
   4. Multiple myeloma.
   5. Solid organ transplant.
   6. History of severe hepatic disease/liver transplant/pending liver transplant.

Ages: 40 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Cancer detection rate (CDR) | Up to 1 year
  The CDR is defined as the number of breast cancers identified per 1,000 magnetic resonance imaging (MRI) screening examinations performed 1 year following supplemental screening MRI.

SECONDARY OUTCOMES:
CDR of participants designated as low risk using the Tyrer-Cuzick (TC) criteria | Up to 1 year
  Cancer detection rate is defined as the number of breast cancers identified per 1,000 MRI screening examinations performed of supplemental screening breast MRI in participants with high Mirai risk and low (<20%) lifetime TC risk.
Comparison of CDR in low and high TC risk groups | Up to 1 year
  The CDR of supplemental screening breast MRI in participants with high Mirai risk and high (≥ 20%) lifetime TC risk versus CDR in participants with high Mirai risk and low (<20%) lifetime TC risk will be compared using a two-proportion exact test.
Positive predictive value of supplemental MRI screening and BI-RADS Score (PPV1) | Up to 1 year
  PPV1 is the percentage of all positive supplemental MRI screening in participants with high Mirai risk (Breast Imaging Reporting and Data System (BI-RADS) 3, 4, or 5) for which the participant was found to be positive for cancer within 1 year from the time of MRI.
Positive predictive value of supplemental MRI screening recommending histological or surgical follow-up (PPV2) | Up to 1 year
  PPV2 is the percentage of all supplemental MRI screenings in participants with high Mirai risk recommended for tissue diagnosis or surgical consultation (BI-RADS 4 and 5) that resulted in a histological diagnosis of cancer within 1 year.
Positive predictive value of biopsies resulting in histological diagnosis (PPV3) | Up to 1 year
  PPV3 is the percentage of all known biopsies performed as a result of positive supplemental MRI screening (BI-RADS 4 or 5) that resulted in a tissue diagnosis of cancer within 1 year.
False Positive Rate (FPR) | Up to 1 year
  A false positive is defined as an imaging result that incorrectly identifies a condition as present. The FPR = (False Positives / Total Tests) × 100 (or 1 - specificity) of results on supplemental screening MRIs in participants with high Mirai risk.
Mean tumor size detected in supplemental imaging | Up to 1 year
  Mean tumor size in millimeters (mm) with in situ and invasive components separately on supplemental screening MRI in Mirai high risk participants.
Frequency of tumor stage detected in supplemental imaging | Up to 1 year
  The frequency of tumor stage diagnosed using the supplemental screening MRI in Mirai high risk participants will be reported.
Proportion of participants with Ki-67 expressed biomarker | Up to 1 year
  Ki-67 is divided according to percentage levels: < 15% and > 15%. The proportion of participants with pathologically confirmed Ki-67 by percentage level will be reported.
Proportion of participants with lymph node involvement detected in supplemental imaging | Up to 1 year
  The proportion of participants with demonstrated lymph node involvement of cancers detected on the supplemental screening MRI in Mirai high risk participants.
Correlation between race/ethnicity and CDR | Up to 1 year
  The Spearman's correlation coefficient (rs) will be used to measure the strength and direction of association between race/ethnicity and CDR. The Spearman correlation coefficient, rs, results in values from +1 to -1 where a value of +1 indicates a perfect association, and rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association
Correlation between menopausal status and CDR | Up to 1 year
  The Spearman's correlation coefficient (rs) will be used to measure the strength and direction of association between menopausal status and CDR. The Spearman correlation coefficient, rs, results in values from +1 to -1 where a value of +1 indicates a perfect association, and rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association
Correlation between hormonal status and CDR | Up to 1 year
  The Spearman's correlation coefficient (rs) will be used to measure the strength and direction of association between hormonal status and CDR. The Spearman correlation coefficient, rs, results in values from +1 to -1 where a value of +1 indicates a perfect association, and rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association.
Correlation between breast density and CDR | Up to 1 year
  The Pearson correlation coefficient (r) will be used to measure the strength and direction of association between breast density and CDR. The Pearson correlation coefficient (r) can take values from +1 to -1 where a value of +1 indicates a perfect association, a value of 0 indicates no association, and a value of -1 indicates a perfect negative association. The closer r is to 0, the weaker the association.
Correlation between family history of cancer and CDR | Up to 1 year
  The Spearman's correlation coefficient (rs) will be used to measure the strength and direction of association between history of cancer and CDR. The Spearman correlation coefficient, rs, results in values from +1 to -1 where a value of +1 indicates a perfect association, and rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Chung, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with research collaborators during the course of the study.
Supporting Information: Study Protocol, SAP, ICF